CLINICAL TRIAL: NCT05932316
Title: Evaluating Bronchodilator Response in Patients With Bronchiectasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Mordechai Pollak MD, MSc, Dr Mordechai Pollak, Rambam Health Care Campus
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 0025-23-RMB
Record Dates: First submitted 2023-05-31; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Bronchiectasis; Cystic Fibrosis; Primary Ciliary Dyskinesia; Primary Immune Deficiency; Bronchiolitis Obliterans
Keywords: Bronchodilator response
MeSH Terms: conditions — Bronchiectasis; Cystic Fibrosis; Ciliary Motility Disorders; Primary Immunodeficiency Diseases; Bronchiolitis Obliterans | interventions — Spirometry; Respiratory Function Tests; Albuterol; Bronchodilator Agents

STUDY DESIGN:
Intervention Model Description: Each group of patients and controls will be randomly assigned to two study arms as follows: patients in both arms will perform regular spirometry. After the first series of spirometry testing, patients in the first arm will receive bronchodilators as per bronchodilator response protocol (Salbutamol, 100 mcg, 4 puffs via spacer) and patients in the second arm will receive four puffs of placebo. After a waiting time of 15 minutes, spirometry will be repeated. Following the second spirometry testing those who received salbutamol will now receive placebo and those receiving placebo will receive Salbutamol. After a second period of 15 minutes, a third series of spirometry will be recorded.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The Salbutamol inhaler and the placebo inhaler will be marked as '1' and '2'. The division Nurse will be in charge of marking the inhalers and all the rest of the team and participants will be blinded. The clinicians, technicians and patients will not be able to distinguish between Salbutamol and placebo, and will not know to what arm the patient was assigned at the time of the testing and the interpretation of the results.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Salbutamol first (Other): Individuals included in this arm will receive 4 puffs of Salbutamol prior to the second set of spirometry testing, and 4 puffs of Placebo prior to the third set of spirometry.
  Interventions: Diagnostic Test: spirometry; Drug: Salbutamol; Drug: placebo
- Placebo First (Other): Individuals included in this arm will receive 4 puffs of placebo prior to the second set of spirometry testing and 4 puffs of Salbutamol prior to the third set of spirometry testing.
  Interventions: Diagnostic Test: spirometry; Drug: Salbutamol; Drug: placebo

INTERVENTIONS:
Diagnostic Test: spirometry — participants will undertake spirometry testing before and after bronchodilators and placebo
  Other Names: pulmonary function testing
Drug: Salbutamol — Salbutamol inhalation to determine bronchodilator response
  Other Names: bronchodilator
Drug: placebo — placebo inhalation prior to repeating spirometry

SUMMARY:
Although patients with bronchiectasis tend to have non reversible obstructive patterns on pulmonary function tests (PFTs), reversible obstruction is not uncommon. While bronchodilator response (BDR) is a main characteristic of asthma, the pathophysiology causing this phenomenon in bronchiectasis patients is less clear.

The goal of this clinical trial is to assess BDR in patients with bronchiectasis.

The main aims of this study:

1. To evaluate the role of bronchodilators in BDR testing of patients with bronchiectasis.
2. Characterize and compare BDR between different subgroups of patients with bronchiectasis, and compared to patients without bronchiectasis (healthy controls).
3. Identify demographics and other clinical variables associated with positive BDR

Participants will be taking a series of three spirometry tests: After the first spirometry testing, patients will be randomly assigned to receive bronchodilators as per bronchodilator response protocol (Salbutamol, 100 mcg, 4 puffs via spacer) or four puffs of placebo. After a waiting time of 15 minutes, spirometry will be repeated. Following the second spirometry testing those who received salbutamol will now receive placebo and those receiving placebo will receive Salbutamol. After a second period of 15 minutes, a third series of spirometry will be recorded.

DETAILED DESCRIPTION:
Bronchiectasis are defined as irreversible dilatation of the bronchial tree. Patients with bronchiectasis suffer of chronic cough and sputum production, and are predisposed to recurrent airway infections. Many systemic diseases can cause bronchiectasis: cystic fibrosis (CF), primary ciliary dyskinesia (PCD), primary immune deficiencies (PID) and idiopathic bronchiectasis (IB) represent a significant proportion of patients with bronchiectasis starting in early age.

Pulmonary function testing (PFT) and specifically forced expiratory volume in one second (FEV1) is a common modality used to estimate lung disease progression and pulmonary exacerbations in patients with bronchiectasis. Although patients with bronchiectasis tend to have non reversible obstructive patterns on pulmonary function tests (PFTs), reversible obstruction is not uncommon. While bronchodilator response (BDR) is a main characteristic of asthma, the pathophysiology causing this phenomenon in bronchiectasis patients is less clear. The improvement in FEV1 after inhalation of bronchodilators can be attributed to bronchodilation or improved mucociliary clearance. It can be speculated that for some of the bronchiectasis patients, hyper-reactive airways or asthma can contribute to the reversible pattern. Despite the wide scale use of bronchodilators in bronchiectasis the evidence for its efficacy is lacking. While some studies found that BDR is associated with more severe disease, other studies did not find such associations.

According to ATS/ERS statement, the proper way to determine BDR, is by first recording three attempts of spirometry, then delivering bronchodilators, and after a waiting time, obtaining again at least three attempts of spirometry. The most resent ATS/ERS technical standard suggests that change of >10% relative to the predicted value for FEV1 or forced vital capacity (FVC) be considered a positive BDR.

While in most scenarios it is reasonable to assume that the change in FEV1 measured after the waiting time can be attributed solely to the affect of bronchodilators, this is not necessarily the case in bronchiectatic diseases. Theoretically, in bronchiectasis, the forced expiration maneuver used in spirometry testing can potentially cause changes in lung function, for example by inducing cough and mobilization of sputum. Evidence for this assumption can be seen in that respiratory therapy in terms if positive expiratory pressure (PEP) therapy can improve various parameters of lung function when tested again closely after the therapy.

The goal of this study is to determine if bronchodilator response in bronchiectatic disease might be influenced by other factors apart from the direct effect of bronchodilators. Secondary objectives are to assess if BDR is associated with age, gender, specific bronchiectatic disease, baseline FEV1, and other clinical factors such as sputum cultures, IgE levels, eosinophil levels, computed tomography (CT) score, family history of asthma and use of inhaled steroids.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bronchiectasis confirmed by CT scan
* No recent pulmonary exacerbation as determined by prescription of systemic antibiotics in 7 days prior to BDR testing
* No use of long-acting beta agonists (LABA) 12 hours before BDR testing or short acting beta agonist (SABA) 4 hours before testing

Exclusion Criteria:

* Patients under 5 years of age
* Patients incapable to perform proper spirometry

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Bronchodilator response compared to placebo (change in FEV1) | spirometry results will be collected in one clinic visit in three steps: *baseline *15 minutes after first intervention (placebo or salbutamol) *15 minutes after second intervention (placebo or salbutamol)
  Bronchodilator response = change in forced expiratory volume 1 second (FEV1) from pre to post salbutamol inhalation, compared to the same change after placebo. Results will be presented in "percent predicted" using global lung initiative (GLI) equations.
Bronchodilator response compared to placebo (change in FVC) | spirometry results will be collected in one clinic visit in three steps: *baseline *15 minutes after first intervention (placebo or salbutamol) *15 minutes after second intervention (placebo or salbutamol)
  Bronchodilator response = change in forced vital capacity (FVC) from pre to post salbutamol inhalation, compared to the same change after placebo. Results will be presented in "percent predicted" using global lung initiative (GLI) equations.

SECONDARY OUTCOMES:
response in specific bronchiectatic disease | spirometry results will be collected in one clinic visit in three steps: *baseline *15 minutes after first intervention (placebo or salbutamol) *15 minutes after second intervention (placebo or salbutamol)
  assessment of bronchodilator response (change in forced expiratory volume 1 second (FEV1) from pre to post salbutamol inhalation) differences between different types of bronchiectatic disease (cystic fibrosis (CF), Primary ciliary dyskinesia (PCD), non CF - non PCD bronchiectatic disease) Results will be presented in "percent predicted" using global lung initiative (GLI) equations.
bronchiectasis compared to healthy controls | spirometry results will be collected in one clinic visit in three steps: *baseline *15 minutes after first intervention (placebo or salbutamol) *15 minutes after second intervention (placebo or salbutamol)
  assessment of BDR (change in forced expiratory volume 1 second (FEV1) from pre to post salbutamol inhalation) differences between patients with bronchiectatic disease and healthy controls Results will be presented in "percent predicted" using global lung initiative (GLI) equations.
Bronchodilator response by age | spirometry results will be collected in one clinic visit in three steps: *baseline *15 minutes after first intervention (placebo or salbutamol) *15 minutes after second intervention (placebo or salbutamol)
  Identify if bronchodilator response (change in forced expiratory volume 1 second (FEV1) from pre to post salbutamol inhalation, presented in "percent predicted" using global lung initiative (GLI) equations) is influenced by the age of the participant
Bronchodilator response by sex | spirometry results will be collected in one clinic visit in three steps: *baseline *15 minutes after first intervention (placebo or salbutamol) *15 minutes after second intervention (placebo or salbutamol)
  Identify if bronchodilator response (change in forced expiratory volume 1 second (FEV1) from pre to post salbutamol inhalation, presented in "percent predicted" using global lung initiative (GLI) equations) is influenced by the biological sex of the participant
Bronchodilator response by bronchiectatic disease | spirometry results will be collected in one clinic visit in three steps: *baseline *15 minutes after first intervention (placebo or salbutamol) *15 minutes after second intervention (placebo or salbutamol)
  Identify if bronchodilator response (change in forced expiratory volume 1 second (FEV1) from pre to post salbutamol inhalation, presented in "percent predicted" using global lung initiative (GLI) equations) is influenced by the specific bronchiectatic disease (cystic fibrosis (CF), Primary ciliary dyskinesia (PCD), non CF - non PCD bronchiectatic disease).
Bronchodilator response by use of inhaled steroids | spirometry results will be collected in one clinic visit in three steps: *baseline *15 minutes after first intervention (placebo or salbutamol) *15 minutes after second intervention (placebo or salbutamol)
  Identify if bronchodilator response (change in forced expiratory volume 1 second (FEV1) from pre to post salbutamol inhalation, presented in "percent predicted" using global lung initiative (GLI) equations) is influenced by the use of inhaled corticosteroids.
Bronchodilator response by history of allergy | spirometry results will be collected in one clinic visit in three steps: *baseline *15 minutes after first intervention (placebo or salbutamol) *15 minutes after second intervention (placebo or salbutamol)
  Identify if bronchodilator response (change in forced expiratory volume 1 second (FEV1) from pre to post salbutamol inhalation, presented in "percent predicted" using global lung initiative (GLI) equations) is influenced by personal history of allergy
Bronchodilator response by baseline FEV1 | spirometry results will be collected in one clinic visit in three steps: *baseline *15 minutes after first intervention (placebo or salbutamol) *15 minutes after second intervention (placebo or salbutamol)
  Identify if bronchodilator response (change in forced expiratory volume 1 second (FEV1) from pre to post salbutamol inhalation, presented in "percent predicted" using global lung initiative (GLI) equations) is influenced by baseline FEV1 as determined by the best FEV1 measured in the 6 months prior to the day of the study
Bronchodilator response by history of pseudomonas | spirometry results will be collected in one clinic visit in three steps: *baseline *15 minutes after first intervention (placebo or salbutamol) *15 minutes after second intervention (placebo or salbutamol)
  Identify if bronchodilator response (change in forced expiratory volume 1 second (FEV1) from pre to post salbutamol inhalation, presented in "percent predicted" using global lung initiative (GLI) equations) is influenced by personal history of pseudomonas growing in sputum cultures
Bronchodilator response by bronchiectasis severity | spirometry results will be collected in one clinic visit in three steps: *baseline *15 minutes after first intervention (placebo or salbutamol) *15 minutes after second intervention (placebo or salbutamol)
  Identify if bronchodilator response (change in forced expiratory volume 1 second (FEV1) from pre to post salbutamol inhalation, presented in "percent predicted" using global lung initiative (GLI) equations) is influenced by the severity of bronchiectasis as measured by CT imaging using the Bhalla score

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai Pollak, MD, MSc, Principal Investigator — pediatric pulmonology institute, Ruth Rappaport children's hospital, Rambam medical center
Locations (1):
- Rambam Health Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No